CLINICAL TRIAL: NCT06010446
Title: Intravenous Continuous LMWH (enoxaparin) Seems to Be Safe Alternative to UFH in Patients with VV ECMO
Brief Title: Intravenous Continuous LMWH Seems to Be Safe Alternative to UFH in VV ECMO Patients
Status: Completed | Type: Observational
Sponsor: University Hospital, Motol (Other)
Responsible Party: Principal Investigator, Durila Miroslav MUDr. Ph.D., prof.MD. Miroslav Durila, Ph.D., MHA, University Hospital, Motol
Other Study IDs: 15082023
Record Dates: First submitted 2023-08-15; First posted 2023-08-24 (Actual); Last update posted 2025-02-25 (Actual); Status verified 2025-02

CONDITIONS: Refractory Respiratory Failure
MeSH Terms: conditions — Respiratory Insufficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: No intervention, just retrospective analysis of data.

SUMMARY:
Unfractionated heparin (UFH) is worldwide anticoagulation used and recommended anticoagulation in patients with ECMO support. However, it is accompanied with incidence of bleeding or thrombotic compliaction at about 40-60% and high mortality. Because ECMO produce primary haemosthasis pathology, there is a theory that prophylaxis of thrombosis with low molecular weight heparin (LMWH) e.g. Enoxaparin might be sufficient to prevent ECMO throbosis and thrombosis development in patients.

We decided to performed retrospective observation study and analysis of data, from may 2019 until august 2023, in all patients who were put on VV ECMO and to analysis incidence of bleeding, thrombotic and neurologic complications.

DETAILED DESCRIPTION:
Unfractionated heparin (UFH) is worldwide anticoagulation used and recommended anticoagulation in patients with ECMO support. However, it is accompanied with incidence of bleeding or thrombotic compliaction at about 40-60% and high mortality. Because ECMO produce primary haemosthasis pathology, there is a theory that prophylaxis of thrombosis with low molecular weight heparin (LMWH) e.g. Enoxaparin might be sufficient to prevent ECMO throbosis and thrombosis development in patients. This phenomenon of primary haemosthasis pathology may protect ECMO from thrombotic complication as primary haemosthasis plays major role in haemosthasis taking places in high shear stress condiditon such as ECMO. Because LMWH is connected with lower incidence of bleeding complication and HIT (heparin induced thrombocytopenia) in general, in case that patients on VV ECMO developed primary haemosthasis pathology detected by PFA 200, we started to use LMWH instead of UFH in VV ECMO patients.

We decided to performed retrospective observation study and analysis of data, from may 2019 until august 2023, in all patients who were put on VV ECMO and to analysis incidence of bleeding, thrombotic and neurologic complications. We want to compare this incidence of compliactions with data known from patients with other studies using UFH.

ELIGIBILITY:
Inclusion Criteria:

* VV ECMO - use of 2 separate cannulas (jugular and femoral)
* anticoagulation with only intravenous continuous LMWH (Enoxaparin)
* only a period of the first ECMO set running

Exclusion Criteria:

* pregnancy
* Avalon cannula (one double lumen cannula)
* patients after thoraco-abdominal surgery
* patients after lung transplantation in early postoperative period
* patients after trauma without any type of heparin ,,heparin free" ECMO

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with respiratory failure put VV ECMO
Sampling Method: Non-Probability Sample
Enrollment: 43 (Actual)
Dates: Start 2019-05-15 (Actual); Primary Completion 2023-08-15 (Actual); Study Completion 2023-08-15 (Actual)

PRIMARY OUTCOMES:
Incidence of major bleeding complications | Daty from may 2019 till august 2023
  Defined by ECMO registry
Incidence of major thrombotic complications | Daty from may 2019 till august 2023
  Defined by ECMO registry
Incidence of major neurologic complications | Daty from may 2019 till august 2023
  Defined by ECMO registry

CONTACTS AND LOCATIONS:
Overall Officials: Miroslav Durila, prof., Principal Investigator — Department of anesthesiology and intensive care medicine, Motol Hospital
Locations (1):
- Unoversity Hospital Motol, Department of Anaesthesiology and Intensive Care, Prague, Czechia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Durila M, Vajter J, Garaj M, Berousek J, Lischke R, Hlavacek M, Vymazal T. Intravenous enoxaparin guided by anti-Xa in venovenous extracorporeal membrane oxygenation: A retrospective, single-center study. Artif Organs. 2025 Mar;49(3):486-496. doi: 10.1111/aor.14879. Epub 2024 Oct 3. PMID 39360891